CLINICAL TRIAL: NCT01048476
Title: Effects of Lutein and Zeaxanthin Supplementation on Age-related Macular Degeneration
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Le MA, MAL, Peking University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NSFC30872113
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Age-related Macular Degeneration
Keywords: AMD
MeSH Terms: conditions — Macular Degeneration | interventions — Lutein; Zeaxanthins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group L20 (Active Comparator): Dietary Supplement: 20mg Lutein; daily supplementation one year
  Interventions: Dietary Supplement: lutein
- Group L10 (Active Comparator): Dietary Supplement: 10mg Lutein; daily supplementation one year
  Interventions: Dietary Supplement: Lutein
- Group Placebo (Placebo Comparator): Dietary Supplement: Placebo, 0 mg Lutein
  Interventions: Dietary Supplement: placebo
- Active Comparator: Group LZ (Active Comparator): Dietary Supplement: 10mg Lutein and 10mg zeaxanthin; daily supplementation one year
  Interventions: Drug: Lutein and zeaxanthin

INTERVENTIONS:
Dietary Supplement: lutein — Dietary Supplement: 20mg Lutein; daily supplementation one year
  Arms: Group L20
Dietary Supplement: Lutein — Dietary Supplement: 10mg Lutein; daily supplementation one year
  Arms: Group L10
Dietary Supplement: placebo — Dietary Supplement: placebo; daily supplementation one year
  Arms: Group Placebo
Drug: Lutein and zeaxanthin — Dietary Supplement: 10mg Lutein and 10mg zeaxanthin; daily supplementation one year
  Arms: Active Comparator: Group LZ

SUMMARY:
Lutein is one of oxygenated carotenoids. Over the past few years, there has been increased interest in evaluating the effect of lutein for optimizing eye health. A large number of epidemiological studies support the notion that the high intake dietary of lutein is strongly associated with a decreased relative risk of AMD.Moreover, findings from initial observational studies have now been followed by placebo-controlled intervention trials showing that dietary modification and supplementation with lutein result in increasing the macular pigment optical density, and may help to improve visual function in patients suffering from AMD.Currently, nutritional status and background information of lutein and zeaxanthin in Chinese population is lack. Little is known about the preventive and therapy benefits of lutein on visual function in the AMD populations. In particular, the effect on visual function of relatively certain doses of lutein and zeaxanthin is unknown. Therefore, the objective of the present study was to examine the effect of consuming different doses of lutein on MPOD and visual function in AMD.

DETAILED DESCRIPTION:
We aim to study the effect and the mechanism of lutein in the prevention and treatment for age-related macular degeneration (AMD). Using the cluster sampling method, baseline characteristics screening will be performed in Han nationality men and women in the suburban areas of Beijing, ranging in age from 50 to79 years. According to clinical diagnosis standard of AMD, AMD (n=120) and normal subjects (n=40) will be randomly selected to measure serum lutein and nutritional status, and evaluate the relationship between lutein and AMD. Each subject of AMD will be randomly assigned to 1 of 4 groups: Group low lutein (Group LL); Group high lutein (Group HL); Group lutein/zeaxanthin (Group LZ); and Group Placebo to participate in the randomized, double-blind, placebo-controlled, 1 year intervention study, respectively. Macular pigment optical density,related symptoms and multifocal electroretinogram (mfERG) will be measured at at weeks 0, 24 and 48, to compare their dynamic changes in response to supplements at baseline and each follow-up visit, observe time- and dose-response correlation of supplementation with lutein, assess the efficacy, dosage of lutein and/or zeaxanthin supplement.

ELIGIBILITY:
Inclusion Criteria:

* Patients with nonexudative AMD (either categories 2, 3 or 4 according to the AREDS criteria; in group 4 the eyes with no-advanced AMD will be included)
* Age between 50 and 90 years
* Able to understand and comply with the requirements of the trial
* Visual acuity > 0.4
* Subjects must agree to take only the nutritional supplement that is

Exclusion Criteria:

* Currently enrolled in an ophthalmic clinical trial
* Eyes with concomitant macular or choroidal disorders other than AMD and with indefinite signs of AMD
* Eyes with a diagnosis of exudative AMD with active subretinal neovascularization (SRNV) or CNV lesions requiring laser photocoagulation in the study eye
* Subjects with significant ocular lens opacities causing vision decrease
* Subjects with amblyopia
* Subjects with optic nerve disease (neuropathy, atrophy, papilledema), unstable glaucoma as defined by intraocular pressures greater than 25 mm Hg, 3 or more glaucoma medications, C/D of 0.8 or greater and visual fields consistent with glaucoma; history of retina-vitreous surgery, degenerative myopia, active posterior intraocular inflammatory disease, chronic use of topical ocular steroid medications, vasoproliferative retinopathies (other than AMD), rhegmatogenous retinal detachment, and inherited macular dystrophies
* Subjects with demand type pacemakers or epilepsy
* Subjects with uncontrolled hypertension (defined as diastolic of 90 or greater and systolic of 150 or greater)
* Subjects with recent history (within the previous year) of cerebral vascular disease
* manifested with transient ischemic attacks (TIA's) or cerebral vascular accidents (CVA's)
* Subjects with a history of AIDS
* lutein supplementation within the last 3 months
* Subjects who have had intraocular surgery in trial eye within 3 months prior to enrolling in the trial
* Patients who are unwilling to adhere to visit examination schedules

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-04 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
MPOD and multifocal electroretinograms | 1 year

SECONDARY OUTCOMES:
the safety and efficacy of lutein in reducing the risk of the development of advanced AMD. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Peking university, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Evans JR, Lawrenson JG. Antioxidant vitamin and mineral supplements for slowing the progression of age-related macular degeneration. Cochrane Database Syst Rev. 2023 Sep 13;9(9):CD000254. doi: 10.1002/14651858.CD000254.pub5. PMID 37702300